CLINICAL TRIAL: NCT03853174
Title: Effect of Exercise Training on Inflammatory Mediators in COPD
Brief Title: Exercise Training and Inflammatory Mediators in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Medicine, Sousse (Other)
Responsible Party: Principal Investigator, Acheche Amal, PhD student, Faculty of Medicine, Sousse
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COPD and exercise
Record Dates: First submitted 2019-02-21; First posted 2019-02-25 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: COPD
Keywords: COPD; Inflammation; exercise training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Inflammation | interventions — Endurance Training; Resistance Training

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ET (Active Comparator): Active Comparator: ET Endurance training were prformed. Intensity was gradually increased.
  Interventions: Other: Endurance Training ET
- RT (Other): Resistance training were prformed. Intensity was gradually increased.
  Interventions: Other: Resistance Training RT

INTERVENTIONS:
Other: Endurance Training ET — Endurance training were prformed. Intensity was gradually increased.
  Arms: ET
Other: Resistance Training RT — Resistance training were prformed. Intensity was gradually increased.
  Arms: RT

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is widely spread all over the world. It is predicted to be the third leading cause of death by 2020[1]. COPD is a common, preventable treatable disease that is characterized by an airflow limitation which is not fully reversable[2].

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is widely spread all over the world. It is predicted to be the third leading cause of death by 2020. COPD is a common, preventable treatable disease that is characterized by an airflow limitation which is not fully reversable.Not only the long-term exposition to noxious particles and gases contributes to the development of COPD, but also so many others factors such as genetics and cigarette smoking. It has been shown that cigarettes are harmful and contributed to different extra pulmonary disorders. Indeed, it induced a systemic inflammation that was considered as a key process in the pathogenesis of COPD and triggered the activation of inflammatory cells and an abnormal increase of circulating cytokines such as CRP, interleukin (IL6), IL8, tumor necrosis factor alpha (TNF alpha) and leptin.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosed by pulmonary function testing
* Clinically stable
* Abscence of other obstructive diseases
* Signed written consent

Exclusion Criteria:

* Neuromuscular diseases -Severe psychiatric, neurologic or musculoskeletal conditions and /or instable--- --
* cardiovascular diseases.
* Contre-indications to physical therapy
* Acute exacerbations a month before the intervention

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-04-27 (Actual)

PRIMARY OUTCOMES:
Enzyme linked immunosorbent assay for serum cytokines levels change | Baseline, 6 months
  The interleukines were determined by ELISA assays with commercial kits

CONTACTS AND LOCATIONS:
Overall Officials: Amal Acheche, Phd, Principal Investigator — Faculty of Medicine of Sousse Sousse, Tunisia
Locations (1):
- Amal Acheche, Sousse, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] authors non mentionned., global initiative for chronic lung disease. 2017
- [Background] Molfino NA, Jeffery PK. Chronic obstructive pulmonary disease: histopathology, inflammation and potential therapies. Pulm Pharmacol Ther. 2007;20(5):462-72. doi: 10.1016/j.pupt.2006.04.003. Epub 2006 May 6. PMID 16798034
- [Background] Barnes PJ. Inflammatory mechanisms in patients with chronic obstructive pulmonary disease. J Allergy Clin Immunol. 2016 Jul;138(1):16-27. doi: 10.1016/j.jaci.2016.05.011. Epub 2016 May 27. PMID 27373322
- [Background] Barnes PJ. Cellular and molecular mechanisms of chronic obstructive pulmonary disease. Clin Chest Med. 2014 Mar;35(1):71-86. doi: 10.1016/j.ccm.2013.10.004. Epub 2013 Dec 12. PMID 24507838